CLINICAL TRIAL: NCT04663009
Title: Use of a Load Distributing Band Device Compared With Manual Technique for Out of Hospital Cardiac Arrest Patients on Outcome and Cardiopulmonary Resuscitation Process. A Retrospective Clinical Study.
Brief Title: AutoPulse Compared With Manual Technique for OHCA Patients on Outcome and CPR Process.
Status: Completed | Type: Observational
Sponsor: Lars Wik (Other)
Collaborators: Jon Erik Steen Hansen (Unknown); Unai Irusta Zarandona (Unknown); Elisabete Aramendi (Unknown); Erik Alonso (Unknown); Simone Savastano (Unknown); Enrico Baldi (Unknown); Alessandra Palo (Unknown)
Responsible Party: Sponsor-Investigator, Lars Wik, MD, PhD, Ullevaal University Hospital
Organization: Oslo University Hospital (Other)
Other Study IDs: 11903
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Cardiac Arrest; Out-Of-Hospital Cardiac Arrest
Keywords: survival; rosc; cpr process
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Mechanical chest compression: Patients recieving LDB CPR
  Interventions: Device: AutoPulse
- Manual chest compressions: Patients recieving manual CPR

INTERVENTIONS:
Device: AutoPulse — A band circumflex of the chest that provide chest cage compressions.
  Other Names: LDB
  Groups: Mechanical chest compression

SUMMARY:
The AutoPulse Resuscitation System Model 100 (ZOLL Medical Corporation, Chelmsford, MA, US) ZOLL has been used as a standard treatment for a number of subjects in this trial and granted CE marking for Europe in November of 2003. The AutoPulse device is an automated, portable, battery-powered, load-band-distributing (LDB), chest compression device, which provides chest compressions as an adjunct to performing manual cardiopulmonary resuscitation (CPR). Use of the device is intended to provide consistent chest compressions without interruption to a victim of out-of-hospital cardiac arrest (OOHCA), to reduce the impact of rescuer fatigue due to application of manual CPR, and to enable rescuers to address additional patient needs. In the present study investigators will compare electronic data generated during cardiopulmonary resuscitation stored in the different multimonitores between LDB and manual chest compressions.

DETAILED DESCRIPTION:
Load distributing band (LDB) CPR devices have been developed to improve both the quality and consistency of chest compressions during CPR, as well as lessening the pauses in active compressions.12,19,20 The LDB device has been shown to improve hemodynamics both in a porcine model and in humans, but also lower and higher survival to hospital discharge rates using LDB-CPR compared to M-CPR.21 It is important to emphasize the benefit for early use of the device (within 8 minutes of a cardiac arrest). Analysis also showed an improvement in the benefit ratio for centers which used A-CPR over a prolonged period of time.22 Previous clinical hemodynamic studies have demonstrated increased CPP (20 ± 12 mmHg versus 15 ± 11 mmHg, p < 0.015), peak right atrial pressure (129 ± 32 mmHg versus 83 ± 40 mmHg, p < 0.0001), peak aortic pressure (153 ± 28 mmHg versus 115 ± 42 mmHg, p < 0.0001) when comparing A-CPR to MCPR, respectively.20 Research indicates that increased coronary perfusion pressure improves survival.32 One retrospective review of OOHCA patients found a statistically significant increase in ROSC with LDB-CPR (39%) as compared to M-CPR (29%, p < 0.003)21 and another OOHCA trial documented increased survival to ED when patients were treated with LDB-CPR (29%) compared to M-CPR (19%, p < 0.02).22 In another retrospective historically controlled trial, survival rates were significantly better for patients treated with LDB-CPR compared to M-CPR in episodes of OOHCA when used by rapid response EMS personnel. Overall ROSC was 34.5% for LDB-CPR compared to 20.2% for M-CPR. Survival to hospital admission was improved 20.9% vs. 11.1%, and finally, survival to hospital discharge was improved 9.7% compared to 2.9% for M-CPR. However, no difference was found between the survivors of the two groups with respect to cerebral performance or overall performance categories.23,24 A randomized, controlled trial (RCT) compared LDB-CPR to M-CPR with respect to 4 hour survival following the first recorded emergency call (911). This trial was terminated when no difference was found between the two groups in survival to 4 hours. Worse cerebral performance at hospital discharge was found in the A-CPR group.10 However, it may be the case that this trial had a suboptimal design and significant methodological problems.25,27,28 Finally, the largest RCT, CIRC compared integrated LDB-CPR with high quality M-CPR and found that of 4753 randomized patients, 522 (11.0%) met post enrollment exclusion criteria. Therefore, 2099 (49.6%) received integrated LDB (iLDB)-CPR and 2132 (50.4%) M-CPR. Sustained ROSC (emergency department admittance), 24h survival and hospital discharge (unknown for 12 cases) for iLDB-CPR compared to M-CPR were 600 (28.6%) vs. 689 (32.3%), 456 (21.8%) vs. 532 (25.0%), 196 (9.4%) vs. 233 (11.0%) patients, respectively. The adjusted odds ratio of survival to hospital discharge for iLDB-CPR compared to M-CPR, was 1.06 (95% CI 0.83-1.37), meeting the criteria for equivalence. The 20 min CPR fraction was 80.4% for iLDB-CPR and 80.2% for M-CPR. The authors conclude that compared to high-quality M-CPR, iLDB-CPR resulted in statistically equivalent survival to hospital discharge.

In the present study investigators explore both positive and negative effects of LDB- and M-CPR in standard daily EMS treatment of OOHCA patients.

Knowledge is limited as to the best way to optimize resuscitation of patients with OOHCA. This is evidenced by the low survival rates currently being achieved.2,3,4 As is well evidenced, the early onset of improved circulation during resuscitation results in improved survival rates.32,33,34 Experimental animal studies have indicated improved myocardial blood flow and showed improvement in key pressure measurements including aortic and right atrial peak over M-CPR.12 Upon the addition of epinephrine, LDB-CPR also showed increased cerebral blood flow, a key factor in preserving neurological intactness, as well as improving CPP.12 Experimental animal studies also show improvement in survival to neurological intactness of ACPR over M-CPR.19 It appears that the use of the LDB has been associated with increased end-tidal CO2 (ETCO2, versus M-CPR).38,39,40 In one of the studies, there was also a significant increase in short-term survival over that of M-CPR.39 None of these studies were definitive and did not follow the patients for long term survival but they indicated that LDB may be capable of a real contribution to resuscitative medicine and merited a further, more thorough investigation.38,39,40 Several studies have indicated that higher levels of ETCO2 appeared to be prognostic of ROSC.35,36,37 One trial concluded that monitoring of ETCO2 had potential as a noninvasive indicator of cardiac output during resuscitations attempts and could also serve as a prognostic indicator. This same trial reported that if a patient had initial, average and final ETCO2 readings of 10mmHg, they were able to correctly identify 100% of those patients achieving ROSC with specificities of 74.1%, 90% and 81.4% respectively.36 Another trial concluded that ETCO2 may also have value in determining when to terminate resuscitative efforts.37 Although an RCT was inconclusive as to the benefits of use of the LDB-CPR10; a later trial, a non-randomized, phased observational cohort evaluation, resulted in an increase of survival to hospital discharge from 3% to nearly 10%.23,24 Therefore, it has been hypothesized that timely use of an LDB-CPR to assist in improved circulation could significantly increase survival rates. In 2006, Drs. Lewis and Niemann published an editorial in JAMA, further analyzing the outcomes of these seemingly contradictory studies. While indicating that M-CPR may be better than generally recognized, they also state that there are numerous reasons for conflicting results. They agree that it is not possible to reach any definitive conclusions as to the value of LDB-CPR without further investigation. They advocate a well-controlled trial with clearly defined endpoints, with particular mention made of ensuring the quality of M-CPR used as a comparison. Several sources have discussed the many factors that could have influenced outcome, including strong preconceived notions regarding effective therapies as well as factors such as the Hawthorne Effect.25,27,28,41 Drs. Lewis and Niemann said it best when they conclude that "only by aggressively identifying and rigorously testing promising new therapies will the outcome improve for patients who experience sudden cardiac death."25 The CIRC trial was designed with the goal of being such a trial. The goal of that trial was to test the positive results of the non-randomized trial in the context of an RCT, utilizing a protocol designed to determine whether LDB-CPR was superior, or equivalent to M-CPR using evidence-based medical methodologies. The Circulation-Improving Resuscitation Care (CIRC) trial, an international, multi-center trial, was designed to compare the effectiveness of integrated resuscitation (iLDB-CPR) protocol, to conventional M-CPR for the treatment of OOHCA-PCE. Compared to high-quality M-CPR, iLDB-CPR resulted in statistically equivalent survival to hospital discharge.

The investigators are not aware of any previous publication comparing LDB- with M-CPR in a standard OOHCA situation between two different EMS's in respect to outcome and CPR process.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or more (or local age of consent) who suffer arrest of all etiologies in an out-of-hospital setting and who do not meet any of the exclusion criteria below.

Exclusion Criteria:

* Patients must not fulfill any of the following exclusion criteria (See Section 4.2):

  * Wards of the state
  * Prisoner
  * Do Not Attempt to Resuscitate (DNAR) orders
  * Patients whose chest circumference is too big (> 130 cm)
  * Patients whose chest circumference is too small (< 75 cm)
  * Patients whose weight is greater than 150 Kg.
  * CPR device other than LDB device.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in cardiac arrest treated by the EMS at the different sites.
Sampling Method: Probability Sample
Enrollment: 3250 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Survival | through study completion, an average of 1 year
  The primary endpoint is OOHCA patient survival to hospital discharge

SECONDARY OUTCOMES:
Short time survival | through study completion, an average of 1 year
  sROSC and tROSC 24 hours (from time of emergency call) Hospital discharge with Cerebral Performance Category (CPC) 1-2 sROSC and Survival to hospital discharge in the different Utstein categories.
CPR process outcomes | through study completion, an average of 1 year
  Detailed description of delivered shocks related to:
  Chest compressions Chest compression pauses Chest compression cycle Chest compression pre-, post-, peri-shock pauses The total number of defibrillation shocks Time to first shock The duration of pulselessness (from emergency call received to sROSC) Hands-on interval Abrupt stops of chest compression Ventilation during chest compressions and chest compression pause The possible role of the presence of chest compressions artefact on ETCO2 curve on ROSC and survival.
  Comparison of ETCO2 pre and post LDB deployment and its role on ROSC and survival

CONTACTS AND LOCATIONS:
Overall Officials: Lars Wik, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Central Hospital Vestfold, Tønsberg, Norway

IPD SHARING:
Plan to Share IPD: No